CLINICAL TRIAL: NCT02531477
Title: Intra-carotid Anesthetic Agent Delivery
Acronym: ICAAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2
Record Dates: First submitted 2015-07-15; First posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental group (Experimental): Intracarotid injection of propofol to detect efficacy and safety as a novel route for drug delivery
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — intracarotid propofol as an anesthetic agent

SUMMARY:
Intra-Carotid delivery of propofol.

DETAILED DESCRIPTION:
Propofol injection into carotid artery . detection of response of experimental subjects to pain

ELIGIBILITY:
Inclusion Criteria:

* 5 experimental animals (rabbits)

Exclusion Criteria:

* none

Ages: 10 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
effect on painful stimulus perception on HR measurement | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt